**Cover Page** - Study Title: Risk of Anemia Development and Clinical Effects of Oral Iron Therapy in Women (18–55 Years) With Non-Anemic Iron Deficiency - NCT Number: [To be assigned] - Document Date: October 28, 2025

## **Informed Consent Form (English Version)**

**Study Site:** Kağıthane No. 5 Family Health Center (ASM), Çeliktepe, Sarıgöl Cad. Aydınlar Cami Altı No:39 D. 34413 Kağıthane/Istanbul, Turkey

**Study Title:** Risk of Anemia Development and Clinical Effects of Oral Iron Therapy in Women (18–55 Years) With Non-Anemic Iron Deficiency – Medical Specialty Thesis Study

**Purpose of the Study:** Non-anemic iron deficiency is common worldwide. Iron deficiency without anemia (IDWA) may cause fatigue, reduced exercise capacity, and concentration difficulties. Early correction of iron deficiency may improve patient symptoms and quality of life. Evidence regarding iron supplementation in non-anemic individuals is variable, and excessive iron can be harmful.

This study evaluates whether dietary interventions to increase iron intake can prevent progression of iron deficiency to anemia and assesses the effects of oral iron therapy on patient symptoms.

**Study Duration:** 3–4 months per participant; total study duration 6 months.

**Study Procedures:** - Conducted at Kağıthane No. 5 Family Health Center under Dr. Ayşen Fenercioğlu and Dr. Osman Demir. - 60 volunteers meeting criteria will be enrolled. - Blood samples (CBC, biochemistry) collected by trained nurses and analyzed in authorized laboratories. - Participants receive dietary counseling to increase iron intake and absorption (e.g., limiting tea/coffee, reducing antacid use). - Biweekly phone follow-ups monitor health changes; participants not meeting criteria will be withdrawn. - After 2 months, participants are stratified by iron deficiency status; those with persistent deficiency receive 80 mg oral ferrous sulfate for 1 month.

**Possible Risks and Discomforts:** - Mild symptoms during 2-month observation (fatigue, weakness, reduced exercise tolerance, concentration difficulties). - Oral iron therapy may cause nausea, vomiting, indigestion, constipation, diarrhea, or dark stool. - Regular monitoring ensures safety; necessary medical interventions provided.

**Confidentiality:** - Personal information is confidential and used only for research purposes. - Only authorized personnel (ethics committee, inspectors) may access data under confidentiality rules.

**Voluntary Participation:** - Participation is voluntary; withdrawal possible without affecting medical care. - No payment provided; no financial responsibility required.

**Consent:** I have read and understood the information. I had the opportunity to ask questions and received satisfactory answers. I voluntarily agree to participate.

**Permission to Use Data:** - I allow my data to be used in this study. - I allow my data to be used in future related research. - I do not allow my data to be used in any research (if selected).

| <b>Signatures:</b> Participant Name: | Signature: | . Date: |
|--------------------------------------|------------|---------|
|--------------------------------------|------------|---------|

| Person Obtaining Consent Name: Signature: I | Date: |
|---------------------------------------------|-------|
| Witness Name: Signature: Date: | |

Contact Information for Questions or Problems: Dr. Osman Demir – +90 532 291 4470